CLINICAL TRIAL: NCT02840591
Title: A Feasibility Study of Ramelteon and Citicoline for Delirium in a General Inpatient Hospital Population
Brief Title: Ramelteon and Citicoline for Delirium
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped the study due to feasibility issues, no enrollment has taken place.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sherwood Brown, Professor, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 042016-063
Record Dates: First submitted 2016-07-15; First posted 2016-07-21 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Delirium
Keywords: Citicoline, Ramelteon, Rozerem
MeSH Terms: conditions — Delirium | interventions — ramelteon; Cytidine Diphosphate Choline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug Treatment (Experimental): * First 5 consecutive subjects: Ramelteon 8 mg daily at 8 pm for 5 days
  * Next 5 consecutive subjects: Citicoline 250 mg daily at 8 pm for 2 days, followed by citicoline 500 mg daily at 8 pm for 3 days
  * All subjects: Standard medical care
  Interventions: Drug: Ramelteon; Drug: Citicoline
- Observation-Only (No Intervention): Standard medical care

INTERVENTIONS:
Drug: Ramelteon
  Other Names: Rozerem
  Arms: Drug Treatment
Drug: Citicoline
  Arms: Drug Treatment

SUMMARY:
Primary aim of this study is to assess the feasibility of conducting clinical research for delirium (confusion due to medical problems) at Clements University Hospital in Dallas, Texas. A secondary aim is to assess whether an FDA-approved sleeping aid called Ramelteon or an over-the-counter supplement called Citicoline are safe and beneficial in delirium.

DETAILED DESCRIPTION:
This will be a 5-day, non-randomized, open-label, consecutive case series of ramelteon treatment followed by a separate consecutive case series of citicoline treatment, both running in parallel with a non-randomized, observation-only, treatment as usual arm in hospitalized patients with delirium.

On the drug treatment arm, first five consecutive subjects meeting Diagnostic and Statistical Manual (DSM)-5 criteria for delirium will be given ramelteon 8 mg daily at bedtime for 5 days. The next five consecutive patients will be given citicoline 250 mg daily at bedtime for 2 days, followed by 500 mg daily at bedtime for 3 days. Patients on the observation-only arm will be screened and followed similarly, except they will not be given any experimental drugs. All subjects will continue to receive standard medical care for delirium, including optimal medical treatment, psychotropic medications and consultations with specialty services as necessary.

The study is a small pilot to see if there is good feasibility, tolerability and a signal for delirium improvement efficacy with the two medications. The goal is to develop the ability to conduct delirium research at this institution and obtain some preliminary pilot data. These data will be used to design and obtain funding for future, larger research studies. the data from each medication will be examined to look for patterns suggesting that one may be preferable for further research. However, given the very small sample size, meaningful between-group statistical analyses are not possible.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to inpatient units commonly known as 12-South or 12-North at Clements University Hospital
* Has capacity to give informed consent OR legally authorized representative is available at bedside
* Expected duration of hospitalization longer than 48 hours
* Fluent in English
* Can be screened by study physician within 24 hours of admission

Exclusion Criteria:

* History of angioedema or any other allergic reaction with previous ramelteon therapy
* Pregnant or currently breast-feeding
* Concurrent use of fluvoxamine
* Severe hepatic impairment
* Severe obstructive sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Number diagnosed and treated | End of study (anticipated 12 months from beginning of study)
  Number of subjects in each arm that are diagnosed with delirium and treated according to protocol. This is a feasibility measure, the investigators are measuring whether it is possible to screen, enroll, diagnose, treat and monitor a sufficient number of subjects with delirium at the study site.

SECONDARY OUTCOMES:
Frequency of serious, less serious, and minor adverse events as measured by a clinical interview aided by an adverse event checklist | Daily for 5 days
Delirium prevalence | Baseline (Day 0)
  Number of subjects diagnosed with delirium according to Diagnostic and Statistical Manual (DSM)-5 criteria

OTHER OUTCOMES:
Delirium severity | Daily for 5 days
  Score on Delirium Rating Scale-Revised (DRS-R98)
Delirium duration | Daily for 5 days
  Number of days a subject continues to fulfill criteria for DSM-5 delirium diagnosis
Length of hospital stay | through study completion, an average of 1 year
  Measured in days

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No